CLINICAL TRIAL: NCT07000578
Title: The Effect of Hip Joint Orthotic Intervention and Conventional Exercise Training on Spasticity, Balance and Walking Performance in Children With Cerebral Palsy: A Clinical Study
Brief Title: The Effect of Hip Joint Orthotic Intervention and Conventional Exercise Training on Spasticity, Balance and Walking Performance in Children With Cerebral Palsy
Status: Enrolling by invitation | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Demet Sarıyıldız, PhD(c), Principal Investigator, Medipol University
Other Study IDs: E-10840098-202.3.02-2974
Record Dates: First submitted 2025-05-24; First posted 2025-06-03 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Palsy (CP)
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral palsy (SP) is defined as a group of persistent disorders that cause activity limitation of movement and postural development. Children with cerebral palsy are typically born with a normal anatomical hip sequence. The incidence of hip dysplasia reported in patients with cerebral palsy ranges from 2% to 75%. Various non-surgical measures have been used to prevent or slow the progression of spastic hip dysplasia. The therapy program should include activities designed to sustain hip movement and promote weight bearing. However, there is no convincing evidence that treatment alone prevents hip subluxation. To prevent the progression of hip dysplasia, the physical therapy program should include activities designed to increase the functionality of the buttocks and promote weight bearing. In our study, standing strategies will be applied as conventional therapy. Orthotizing, corrective dynamic elastomeric fabric orthoses and taping applications are often used to prevent hip dysplasia. In our study, TheraTogs orthotic garment part, auxiliary dynamic belt material supporting muscles Tog-Rite will be used.Tog-Rite with a width of 7 cm will be made by applying approximately 50-60% stretch with spiral winding from the hip to the bottom of the knee. Positioning will be taught to families and instructed to wear 4 hours a day. Reminders will be made via remote weekly message, families will be able to reach the therapist at any time. Conventional therapy will continue for 2 sessions per week, 45 minutes in a clinical setting. T0: initial assessment, T1: 3ay conventional therapy, T3: 3 months of conventional therapy + positioning with spasticity, balance and impact on walking will be examined. Socia-demographic information forms of the children taken to the study will be recorded. According to the Gross Motor Function Classification System, children of the GMFCS I- II- III level will be taken to work. Children's independence levels will be determined and recorded with the Functional Independence Measure (WeeFIM). Muscle tone will be assessed by the Modified Ashworth Scale. The Pediatric Berg Balance Scale will be applied for functional balance. Balance measurement will be done with the Becure Balance System. Assessment of the gait will be done through the Gillette functional assessment questionnaire. The walking speed will be done with a 10 meter walking test.

ELIGIBILITY:
Inclusion Criteria:

* 4 -16 age range
* Diagnosis of unilateral or bilateral spastic cerebral palsy
* With a tendency to increase in hip muscle imbalance or hip adduction
* At least 10 meters walkable (with independent or auxiliary device)
* GMFCS I- II- III level according to the gross motor function classification system

Exclusion Criteria:

* The presence of dysplasia of the hip
* Severe adductor spasticity, Modified Ashworth Scale ≥ 3
* Botulinum toxin injection into lower extremities in the last 6 months
* Use of drugs to reduce spasticity
* The presence of epilepsy
* Mental inadequacy at a level that cannot understand commands

Ages: 4 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Children with cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | From enrollment to the end of treatment at treatment in 0, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Devrim Tarakcı, Assoc. Dr., Principal Investigator — İstanbul Medipol University
Locations (1):
- İstanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)